CLINICAL TRIAL: NCT02249884
Title: Use of Chamomilla Recutita Gel and Urea Cream to Prevent and Treat Radiodermatitis: Phase 2 Study
Brief Title: Dose-Response Curve: Interventions to Prevent and Treat Radiodermatitis
Acronym: DRCPTR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Brasilia (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Elaine Barros Ferreira, RN, University of Brasilia, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: DRCradiodermatitis
Record Dates: First submitted 2014-09-20; First posted 2014-09-26 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Radiodermatitis
Keywords: radiodermatitis; head and neck neoplasms; Breast Neoplasms; Urea; Matricaria; chamomilla; chamomile
MeSH Terms: conditions — Radiodermatitis; Head and Neck Neoplasms; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Urea Dose A (Experimental): Topical application of the urea cream in concentration A. The product should be applied on the skin three times daily over 3 weeks.
  Interventions: Drug: Urea Dose A
- Urea Dose B (Experimental): Topical application of the urea cream in concentration B. The product should be applied on the skin three times daily over 3 weeks.
  Interventions: Drug: Urea Dose B
- Urea Dose C (Experimental): Topical application of the urea cream in concentration C. The product should be applied on the skin three times daily over 3 weeks.
  Interventions: Drug: Urea Dose C
- Chamomile Dose A (Experimental): Topical application of chamomile recutita gel in concentration A. The product should be applied on the skin three times daily over 3 weeks.
  Interventions: Drug: Chamomile Dose A
- Chamomile Dose B (Experimental): Topical application of chamomile recutita gel in concentration B. The product should be applied on the skin three times daily over 3 weeks.
  Interventions: Drug: Chamomile Dose B
- Chamomile Dose C (Experimental): Topical application of chamomile recutita gel in concentration C. The product should be applied on the skin three times daily over 3 weeks.
  Interventions: Drug: Chamomile Dose C

INTERVENTIONS:
Drug: Urea Dose A — Urea cream for topical use.
  Other Names: Urea cream
  Arms: Urea Dose A
Drug: Urea Dose B — Urea cream for topical use.
  Other Names: Urea cream
  Arms: Urea Dose B
Drug: Urea Dose C — Urea cream for topical use.
  Other Names: Urea cream.
  Arms: Urea Dose C
Drug: Chamomile Dose A — Chamomile gel for topical use.
  Other Names: Chamomile gel
  Arms: Chamomile Dose A
Drug: Chamomile Dose B — Chamomile gel for topical use.
  Other Names: Chamomile gel
  Arms: Chamomile Dose B
Drug: Chamomile Dose C — Chamomile gel for topical use.
  Other Names: Chamomile gel
  Arms: Chamomile Dose C

SUMMARY:
Dose response curve to define the security and tolerable dose to be used for prevention and treatment of radiodermatitis in patients with breast or head and neck cancer.

DETAILED DESCRIPTION:
The study is being conducted in Center for High Complexity Oncology (CACON) located at the University Hospital of Brasília (HUB). Has as its target population subjects diagnosed with breast and head and neck cancer undergoing radiotherapy. Three doses of urea cream are being tested. Participants are subjected to simple randomization technique, in which the members of the study are directly allocated in groups set forth, without any intermediate step. Patients are identified, go to a nursing consultation for general orientations about treatment. After the consultation, patients are invited to participate in the study. The patient should express its acceptance through the informed consent form. Data are being collected through interviews and medical records. Patients are being evaluated during three weeks, considering the toxicity of the intervention and the beginning of radiodermatitis. To evaluate the skin reaction will be applied scale of the Radiation Therapy Oncology Group (RTOG) - Acute Radiation Morbidity Scoring Criteria, Common Terminology Criteria for Adverse Events (CTCAE) and Radiation-Induced Skin Reaction Assessment Scale (RISRAS). For reliable assessment and record of the evolution throughout the treatment and study, patients will be photographed weekly (D0, D5, D10, D15). Will be photographed major regions subject to evaluation: frontal, right side profile and left side profile with Photographic camera Nikon P510. The data will be inserted into Statistical Package for Social Sciences (SPSS), version 18.0, for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Being an adult, over the age of 18 years old
* Owning diagnosis of breast or head and neck cancer
* Being first referred to the radiotherapy protocol
* Have absence of radiodermatitis and integrates skin to start radiotherapy
* Not have presented anticipated reaction of hypersensitivity to chamomile or any plant of the family Asteraceae or Compositae or urea.
* Demonstrate conditions to continue the intervention in their home environment when needed.

Exclusion Criteria:

* Medical prescription for the procedure of data collection, some kind of intervention to prevent radiodermatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Time of occurrence of Radiodermatitis | 3 weeks
  Time of occurrence of Radiodermatitis according with the Radiation Therapy Oncology Group (RTOG).

SECONDARY OUTCOMES:
Indicators of toxicity | 3 weeks
  Evaluate the tolerance and safety of the intervention according to the assessment of toxicity during the intervention.
  To evaluate the toxicity will be considered signs and symptoms referable to the region of application of the product, such as skin rash, urticaria, vesicles, blisters, pustules, as well as the patient's report of discomfort, burning, stinging and itching.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Elaine D Reis, RN PhD, Study Director — University of Brasilia; Marcia A Ciol, PhD, Study Director — University of Washington
Locations (1):
- University Hospital of Brasília, Brasília, Federal District, Brazil